CLINICAL TRIAL: NCT05981365
Title: A Phase 1, Open-Label, Two-Part, Fixed-Sequence, Drug-Drug Interaction Study to Evaluate the Effect of Voxelotor on the Pharmacokinetics of Selected CYP and Transporter Probe Substrates in Healthy Participants
Brief Title: Voxelotor CYP and Transporter Cocktail Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GBT440-0122; C5341029 (Other: Alias Study Number)
Record Dates: First submitted 2023-05-17; First posted 2023-08-08 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Sickle Cell Disease
Keywords: Drug drug interaction
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor; Bupropion; repaglinide; Flurbiprofen; Omeprazole; Midazolam; Metformin; Furosemide; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): To evaluate the effect of multiple doses of voxelotor on the plasma pharmacokinetics (PK) of a single dose of bupropion, repaglinide, flurbiprofen, omeprazole, and midazolam
  Interventions: Drug: Voxelotor; Drug: Bupropion; Drug: Repaglinide; Drug: Flurbiprofen; Drug: Omeprazole; Drug: Midazolam
- Part B (Experimental): To evaluate the effect of multiple doses of voxelotor on the plasma PK of a single dose of metformin, furosemide, and rosuvastatin
  Interventions: Drug: Voxelotor; Drug: Metformin; Drug: Furosemide; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Voxelotor — Drug drug interaction
  Other Names: Oxbryta
Drug: Bupropion — Drug drug interaction
  Other Names: Wellbutrin
  Arms: Part A
Drug: Repaglinide — Drug drug interaction
  Other Names: Prandin
  Arms: Part A
Drug: Flurbiprofen — Drug drug interaction
  Other Names: Ansaid
  Arms: Part A
Drug: Omeprazole — Drug drug interaction
  Other Names: Prilosec
  Arms: Part A
Drug: Midazolam — Drug drug interaction
  Other Names: Dormicum
  Arms: Part A
Drug: Metformin — Drug drug interaction
  Other Names: Glucophage
  Arms: Part B
Drug: Furosemide — Drug drug interaction
  Other Names: Lasix
  Arms: Part B
Drug: Rosuvastatin — Drug drug interaction
  Other Names: Crestor
  Arms: Part B

SUMMARY:
This research study is examining multiple doses of voxelotor (a study drug intended for treatment of sickle cell disease) and how it interacts with additional substrates (substrates are drugs or other substances that are metabolized by cytochrome enzymes. The substrates used in this study are FDA approved medications). The study will help to determine the safety and tolerability of the study drugs taken together, as well as the pharmacokinetics (PK) on how your body processes and responds to the combination of the study drug and substrates. Although these drugs are FDA approved, their use in this study is experimental.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, 2-period evaluation study. This means the study doctor and participants in the study will know what study drugs they are taking. There will be approximately 46 healthy male and female participants between the ages of 18 - 55. There will be two parts of the study: parts A and B.

Part A will consist of 26 healthy male and female participants (at least 20% African American). For Part A, participant involvement is expected to last approximately 81 days, including a 33-day screening period and a 48-day on study period (consisting of 2 study treatment periods, a washout period lasting 7 to 14 days, and the Follow-up visit).

Part B will consist of 20 healthy male and female participants (at least 20% African American). For Part B, participant involvement is expected to last approximately 68 days, including a 33-day screening period and a 35-day on study period (consisting of 2 study treatment periods, a washout period lasting 7 to 14 days, and the Follow-up visit).

You will only be allowed to be in one part of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females ≥ 18 and ≤ 55 years of age inclusive, at the time of signing the informed consent.

  2. No clinically significant findings as assessed by review of medical and surgical history, vital signs assessments, 12-lead electrocardiograms (ECG), physical examination, and clinical laboratory evaluations conducted at screening and day of admission. A single repeat measurement/test may be performed to confirm eligibility based upon initial vital signs, ECG, or clinical laboratory tests abnormalities.

  3. Body mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2, and body weight ≥ 50 kg at screening and Period 1 Day -1. BMI = weight (kg)/(height [m])2

  4. Females of childbearing potential must agree to use a highly effective method of contraception or practice abstinence from 2 weeks prior to study start through 30 days after the last dose of study drug. A highly effective method of contraception is defined as one that results in a low documented failure rate when used consistently and correctly such as: condom plus use of an intrauterine device; intrauterine system or hormonal method of contraception (oral, injected, implanted, or transdermal) for their female partner; or sexual abstinence. Males must be surgically sterilized, or agree to practice true abstinence, or use acceptable contraception if sexually active with a female partner of childbearing potential, throughout the study, and for at least 30 days after the last dose of study drug.

  5. Males must agree not to donate sperm during the study and for 30 days following last dose of study drug.

Exclusion Criteria:

1. Positive pregnancy test or is lactating.
2. History or presence of clinically significant allergic diseases (except for untreated,

   asymptomatic, seasonal allergies) at time of screening in the opinion of the Investigator.
3. History or presence of conditions which, in the opinion of the Investigator, are known to interfere with the absorption, distribution, metabolism, or excretion of drugs, such as previous surgery on the gastrointestinal tract (including removal of parts of the stomach, bowel, liver, or pancreas). Participants who have a history of cholecystectomy and appendectomy are eligible for enrollment.
4. Any signs and/or symptoms of acute illness at screening or Day -1.
5. Abnormal ECG in any of the single ECGs collected at screening or Day -1, including QTcF > 430 msec for males and > 450 msec for females, or any cardiac rhythm other than sinus rhythm that is interpreted by the Investigator to be clinically significant. A single repeat measurement may be performed to re-evaluate ECG abnormalities (ie, to confirm that a participant is eligible). All the single ECGs must be not clinically significant to qualify for enrollment into the study.
6. Resting bradycardia (HR < 45 bpm) or resting tachycardia (HR > 100 bpm) at screening or Day -1. A single repeat measurement may be performed to re-evaluate vital signs abnormalities(ie, to confirm that a participant is ineligible). Each of the readings must be not clinically significant to qualify for enrollment into the study.
7. Hypertension, defined as resting (supine) systolic blood pressure (BP) > 140 mmHg or resting diastolic BP > 90 mmHg at screening or Day -1. A single repeat measurement may be performed to re-evaluate vital signs abnormalities (ie, to confirm that a participant is eligible). Each of the readings must be not clinically significant to qualify for enrollment into the study.
8. Use of prescription medications (with the exception of contraception), any over the counter drugs including herbal preparations including St. John's wort or dietary supplements, or any drugs that induce or inhibit study drug specific CYP450(s) within 14 days or 5 half-lives, whichever is longer, prior to Day -1, or requires continuing use during study participation.
9. Prior exposure to voxelotor/Oxbryta® within the past month.
10. Clinically significant anemia, or has donated blood or blood components exceeding 400 mL within 90 days prior to screening.
11. Positive screen for human immunodeficiency virus 1 (HIV-1) and HIV -2 antibodies, hepatitis A virus antibody, hepatitis B surface antigen, or hepatitis C virus antibody.
12. History or presence of contraindication to the use of midazolam including but not limited to hypersensitivity to benzodiazepines or formulation ingredients, acute narrow-angle glaucoma, myasthenia gravis, severe respiratory insufficiency, or sleep apnea syndrome.
13. Poor CYP2C9 or CYP2C19 metabolizer (determined at screening or available historical data).
14. Participant has an allergy or sensitivity to voxelotor, bupropion, repaglinide, flurbiprofen, omeprazole, or midazolam.

    Part B only
15. History of statin-induced myopathy or serious hypersensitivity reaction to other 3-hydroxy-3-methylglutaryl coenzyme A, reductase inhibitors (statins).
16. Heterozygous or homozygous variant allele carriers of SLCO1B1 (c.521T>C, rs4149056), encoding the hepatic uptake transporter OATP1B1, resulting in decreased transport activity.
17. Participant has an allergy or sensitivity to voxelotor, metformin, furosemide, or rosuvastatin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-0122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 participants (26 in Part A and 18 in Part B) were enrolled in the study.
Groups:
- Part A:Treatment Sequence ABCDEFG: On Day 1 of Period 1, participants were administered a single oral dose of Treatment A (bupropion 150 milligrams [mg], flurbiprofen 50 mg, omeprazole 20 mg, and midazolam 2 mg) and on Day 4, participants received a single oral dose of repaglinide 0.5 mg (Treatment B). Period 1 for Part A was of 5 days. In Period 2, participants were administered once daily oral dose of voxelotor 1500 mg (Treatment C) for 13 days. On Day 2, a single oral dose of bupropion 150 mg (Treatment D) was administered immediately following voxelotor administration. On Day 4, single oral dose of Treatment E (flurbiprofen 50 mg, omeprazole 20 mg and midazolam 2 mg) was administered immediately following voxelotor administration. Participants received Treatment F (single oral dose of repaglinide 0.5 mg) and Treatment G (single oral dose of bupropion 150 mg) on Day 6 and Day 12, immediately following voxelotor administration. Period 2 for Part A was of 15 days. There was a washout period of 7 to 14 days in between Period 1 and 2. Participants had a follow-up visit on Day 28.
- Part B: Treatment Sequence ABCD: On Day 1 of Period 1, participants were administered a single oral dose of Treatment A (metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg). Period 1 for Part B was of 4 days. In Period 2, from Day 1 to Day 3, participants were administered Treatment B (oral doses of voxelotor 1500 mg) orally for 3 days. On Day 4, participants were administered Treatment C (single oral doses of metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg) immediately following voxelotor administration. On Day 5, participants were administered Treatment D (single oral dose of voxelotor 1500 mg). Period 2 for Part B was of 7 days. There was a washout period of 7 to 14 days in between Period 1 and 2. Participants had a follow-up visit on Day 18.
Period: Period 1
Arm/Group | Part A:Treatment Sequence ABCDEFG | Part B: Treatment Sequence ABCD
Started | 26 | 18
Completed | 25 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period
Arm/Group | Part A:Treatment Sequence ABCDEFG | Part B: Treatment Sequence ABCD
Started | 25 | 18
Completed | 25 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Part A:Treatment Sequence ABCDEFG | Part B: Treatment Sequence ABCD
Started | 25 | 18
Completed | 25 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study drug (voxelotor or cocktail drugs [probe substrates]).
Groups:
- Part A:Treatment Sequence ABCDEFG: On Day 1 of Period 1, participants were administered a single oral dose of Treatment A (bupropion 150 mg, flurbiprofen 50 mg, omeprazole 20 mg, and midazolam 2 mg) and on Day 4, participants received a single oral dose of repaglinide 0.5 mg (Treatment B). Period 1 for Part A was of 5 days. In Period 2, participants were administered once daily oral dose of voxelotor 1500 mg (Treatment C) for 13 days. On Day 2, a single oral dose of bupropion 150 mg (Treatment D) was administered immediately following voxelotor administration. On Day 4, single oral dose of Treatment E (flurbiprofen 50 mg, omeprazole 20 mg and midazolam 2 mg) was administered immediately following voxelotor administration. Participants received Treatment F (single oral dose of repaglinide 0.5 mg) and Treatment G (single oral dose of bupropion 150 mg) on Day 6 and Day 12, immediately following voxelotor administration. Period 2 for Part A was of 15 days. There was a washout period of 7 to 14 days in between Period 1 and 2. Participants had a follow-up visit on Day 28.
- Total: Total of all reporting groups
Arm/Group | Part A:Treatment Sequence ABCDEFG | Part B: Treatment Sequence ABCD | Total
Number analyzed (Participants) | 26 | 18 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (8.89) | 36.9 (10.08) | 39.8 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 17 | 13 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 16 | 10 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) for Bupropion
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Period 1 Day 1, Period 2 Day 2 and Period 2 Day 12 for Treatment A, D and G, respectively
Population: Pharmacokinetic (PK) evaluable population included all participants who received at least 1 dose of study drug (voxelotor or cocktail drugs [probe substrates]) and had a sufficient PK profile to derive at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Part A: Period 1: Treatment A: On Period 1 Day 1, participants were administered Treatment A (single oral dose of bupropion 150 mg, flurbiprofen 50 mg, omeprazole 20 mg and midazolam 2 mg).
- Part A: Period 2: Treatment D: On Period 2 Day 2, participants were administered Treatment D (single oral dose of bupropion 150 mg) administered immediately following voxelotor.
- Part A: Period 2: Treatment G: On Period 2 Day 12, participants were administered Treatment G (single oral dose of bupropion 150 mg) administered immediately following voxelotor.
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Nanogram per milliliter (ng/mL) | 160.5 (31) | 201.3 (35) | 191.1 (36)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment D; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.2629, 90% CI 2-sided [1.1673 to 1.3663]
Statistical Analysis 2: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment G; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1845, 95% CI 2-sided [1.0758 to 1.3042]

2. Primary Outcome: Part A: Cmax for Repaglinide
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Period 1 Day 4 and Period 2 Day 6 for Treatment B and F, respectively
Population: PK evaluable population included all participants who received at least 1 dose of study drug (voxelotor or cocktail drugs [probe substrates]) and had a sufficient PK profile to derive at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Part A: Period 1: Treatment B: On Period 1 Day 4, participants were administered a single oral dose of repaglinide 0.5 mg (Treatment B).
- Part A: Period 2: Treatment F: On Period 2 Day 6, participants were administered a single oral dose of repaglinide 0.5 mg (Treatment F) immediately following voxelotor administration.
Arm/Group | Part A: Period 1: Treatment B | Part A: Period 2: Treatment F
Number analyzed (Participants) | 26 | 25
ng/ml | 10.85 (41) | 12.89 (37)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment B vs Part A: Period 2: Treatment F; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1929, 90% CI 2-sided [1.0215 to 1.3930]

3. Primary Outcome: Part A: Cmax for Flurbiprofen
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post-dose on Period 1 Day 1 and Period 2 Day 4 for Treatment A and E, respectively
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Part A: Period 2: Treatment E: On Period 2 Day 4, participants were administered single oral doses of flurbiprofen 50 mg, omeprazole 20 mg, and midazolam 2 mg (Treatment E), immediately following voxelotor administration.
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
ng/ml | 6923 (25) | 7820 (20)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1311, 90% CI 2-sided [1.0496 to 1.2189]

4. Primary Outcome: Part A: Cmax for Omeprazole
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
ng/ml | 458.1 (58) | 374.3 (57)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.8228, 90% CI [0.6992 to 0.9683]

5. Primary Outcome: Part A: Cmax for Midazolam
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
ng/ml | 10.33 (38) | 15.99 (23)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.5738, 90% CI 2-sided [1.4523 to 1.7054]

6. Primary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero (0) to the Time of the Last Quantifiable Concentration (AUCt) for Bupropion
Description: AUCt was calculated using the linear/log trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour* nanogram/milliliter (h*ng/mL)
Groups:
- Part A: Period 1 Treatment A: On Period 1 Day 1, participants were administered Treatment A (single oral dose of bupropion 150 mg, flurbiprofen 50 mg, omeprazole 20 mg and midazolam 2 mg).
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Hour* nanogram/milliliter (h*ng/mL) | 845.3 (29) | 963.9 (28) | 812.1 (28)
Statistical Analysis 1: Comparison: Part A: Period 1 Treatment A vs Part A: Period 2: Treatment D; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1491, 90% CI 2-sided [1.0807 to 1.2220]
Statistical Analysis 2: Comparison: Part A: Period 1 Treatment A vs Part A: Period 2: Treatment G; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.9494, 90% CI 2-sided [0.8759 to 1.0291]

7. Primary Outcome: Part A: AUCt for Repaglinide
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment B | Part A: Period 2: Treatment F
Number analyzed (Participants) | 26 | 25
h*ng/mL | 15.47 (40) | 20.59 (34)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment B vs Part A: Period 2: Treatment F; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.3316, 90% CI 2-sided [1.2558 to 1.4121]

8. Primary Outcome: Part A: AUCt for Flurbiprofen
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 39639 (26) | 44940 (24)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1282, 90% CI 2-sided [1.0700 to 1.1896]

9. Primary Outcome: Part A: AUCt for Omeprazole
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 889.4 (62) | 721.8 (68)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.8047, 90% CI 2-sided [0.7173 to 0.9027]

10. Primary Outcome: Part A: AUCt for Midazolam
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 25.78 (42) | 52.58 (27)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 2.0611, 90% CI 2-sided [1.8789 to 2.2609]

11. Primary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf) for Bupropion
Description: AUCinf was calculated as AUClast + Clast/lamda z, where AUClast: area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration. Clast is the last measurable concentration and lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 1
Population: PK evaluable population included all participants who received at least 1 dose of study drug (voxelotor or cocktail drugs [probe substrates]) and had a sufficient PK profile to derive at least 1 PK parameter. Here "Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 24 | 24
Hour*nanogram/milliliter | 883.3 (30) | 985.4 (28) | 839.1 (28)
Statistical Analysis 1: Comparison: Part A: Period 1 Treatment A vs Part A: Period 2: Treatment G; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1374, 90% CI 2-sided [1.0672 to 1.2122]
Statistical Analysis 2: Comparison: Part A: Period 1 Treatment A vs Part A: Period 2: Treatment G; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.9371, 90% CI 2-sided [0.8643 to 1.0162]

12. Primary Outcome: Part A: AUCinf for Repaglinide
Description: as for outcome 11
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment B | Part A: Period 2: Treatment F
Number analyzed (Participants) | 19 | 20
h*ng/mL | 16.49 (40) | 21.74 (33)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment B vs Part A: Period 2: Treatment F; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.2713, 90% CI 2-sided [1.1939 to 1.3538]

13. Primary Outcome: Part A: AUCinf for Flurbiprofen
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 40047 (26) | 45361 (25)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1270, 90% CI 2-sided [1.0688 to 1.1883]

14. Primary Outcome: Part A: AUCinf for Omeprazole
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 24 | 24
h*ng/mL | 932.3 (62) | 743.1 (69)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.7973, 90% CI 2-sided [0.7039 to 0.9031]

15. Primary Outcome: Part A: AUCinf for Midazolam
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 27.15 (40) | 54.42 (28)
Statistical Analysis 1: Comparison: Part A: Period 1: Treatment A vs Part A: Period 2: Treatment E; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 2.0260, 90% CI 2-sided [1.8496 to 2.2193]

16. Primary Outcome: Part B: Cmax for Metformin
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose on Period 1 Day 1 and Period 2 Day 4 for Treatment A and Treatment C, respectively
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B: Period 1: Treatment A: On Period 1 Day 1, participants were administered single oral doses of metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg (Treatment A).
- Part B: Period 2: Treatment C: On Period 2 Day 4, participants were administered single oral doses of metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg (Treatment C) immediately after a single oral dose of voxelotor 1500 mg.
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
ng/mL | 55.84 (35) | 44.17 (36)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.7909, 90% CI 2-sided [0.7160 to 0.8737]

17. Primary Outcome: Part B: Cmax for Furosemide
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
ng/mL | 48.58 (32) | 52.62 (35)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.0831, 90% CI 2-sided [0.9723 to 1.2065]

18. Primary Outcome: Part B: Cmax for Rosuvastatin
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
ng/mL | 5.545 (46) | 7.286 (53)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.3138, 90% CI 2-sided [1.1871 to 1.4541]

19. Primary Outcome: Part B: AUCt for Metformin
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
h*ng/mL | 303.8 (26) | 241.7 (30)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.7958, 90% CI 2-sided [0.7420 to 0.8534]

20. Primary Outcome: Part B: AUCt for Furosemide
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
h*ng/mL | 105.0 (28) | 108.4 (33)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.0322, 90% CI 2-sided [0.9531 to 1.1179]

21. Primary Outcome: Part B: AUCt for Rosuvastatin
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours post-dose on Day 1 and Day 4 for Treatment A and Treatment C, respectively
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
h*ng/mL | 50.29 (46) | 60.22 (45)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.1975, 90% CI 2-sided [1.0972 to 1.3069]

22. Primary Outcome: Part B: AUCinf for Metformin
Description: as for outcome 11
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
h*ng/mL | 310.5 (25) | 249.0 (29)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 0.8018, 90% CI 2-sided [0.7472 to 0.8604]

23. Primary Outcome: Part B: AUCinf for Furosemide
Description: as for outcome 11
Time Frame: as for outcome 16
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 15 | 17
h*ng/mL | 108.4 (29) | 113.3 (30)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.0630, 90% CI 2-sided [0.9888 to 1.1427]

24. Primary Outcome: Part B: AUCinf for Rosuvastatin
Description: as for outcome 11
Time Frame: as for outcome 16
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 16 | 18
h*ng/mL | 50.87 (45) | 63.16 (43)
Statistical Analysis 1: Comparison: Part B: Period 1: Treatment A vs Part B: Period 2: Treatment C; Analysis was performed using linear mixed model, with treatment as fixed effect and participant as random effect; Test type: Other; Ratio of Geometric LS Means = 1.2197, 90% CI 2-sided [1.1114 to 1.3385]

25. Secondary Outcome: Part A: Cmax for 6-Hydroxybupropion
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
ng/mL | 351.1 (45) | 376.3 (45) | 489.1 (49)

26. Secondary Outcome: Part A: Cmax for 5-Hydroxyomeprazole
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
ng/mL | 179.8 (29) | 216.8 (27)

27. Secondary Outcome: Part A: Cmax for 1-Hydroxymidazolam
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
ng/ml | 5.984 (44) | 7.291 (28)

28. Secondary Outcome: Part A: AUCt for 6-Hydroxybupropion
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
h*ng/mL | 11529 (49) | 11223 (44) | 13453 (53)

29. Secondary Outcome: Part A: AUCt for 5-Hydroxyomeprazole
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 504.1 (21) | 611.4 (21)

30. Secondary Outcome: Part A: AUCt for 1-Hydroxymidazolam
Description: AUCt was calculated using the linear/log trapezoid rule.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 12.73 (43) | 20.07 (27)

31. Secondary Outcome: Part A: AUCinf for 6-Hydroxybupropion
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 19 | 24 | 24
h*ng/mL | 11692 (47) | 12407 (44) | 14990 (55)

32. Secondary Outcome: Part A: AUCinf for 5-Hydroxyomeprazole
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
h*ng/mL | 510.3 (21) | 615.5 (22)

33. Secondary Outcome: Part A: AUCinf for 1-Hydroxymidazolam
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 23 | 25
h*ng/mL | 12.72 (43) | 20.92 (26)

34. Secondary Outcome: Part A: Time at Which Cmax Was Observed (Tmax) for Bupropion
Description: The time that Cmax was observed.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Hours | 1.500 [1.00 to 3.00] | 1.500 [1.00 to 3.00] | 1.500 [1.00 to 3.00]

35. Secondary Outcome: Part A: Tmax for 6-Hydroxybupropion
Description: The time that Cmax was observed for 6-Hydroxybupropion.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Hours | 3.015 [1.13 to 8.05] | 4.000 [2.00 to 8.00] | 3.000 [1.50 to 4.00]

36. Secondary Outcome: Part A: Tmax for Repaglinide
Description: The time that Cmax was observed for Repaglinide.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1: Treatment B | Part A: Period 2: Treatment F
Number analyzed (Participants) | 26 | 25
Hours | 0.500 [0.50 to 1.07] | 0.500 [0.50 to 2.00]

37. Secondary Outcome: Part A: Tmax for Flurbiprofen
Description: The time that Cmax was observed for Flurbiprofen.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 2.000 [0.50 to 6.00] | 1.500 [0.50 to 3.13]

38. Secondary Outcome: Part A: Tmax for Omeprazole
Description: The time that Cmax was observed for Omeprazole.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Groups:
- Part A: Period 1: Treatment A: On Period 1 Day 1, participants were administered single oral doses of metformin hydrochloride 10 mg, furosemide 1 mg, and rosuvastatin 10 mg (Treatment A).
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 3.13]

39. Secondary Outcome: Part A: Tmax for 5-Hydroxyomeprazole
Description: The time that Cmax was observed for 5-Hydroxyomeprazole.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 2.000 [1.00 to 4.02] | 2.000 [1.00 to 4.00]

40. Secondary Outcome: Part A: Tmax for Midazolam
Description: The time that Cmax was observed for Midazolam.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 1.000 [0.50 to 3.00] | 1.000 [0.50 to 1.00]

41. Secondary Outcome: Part A: Tmax for 1-Hydroxymidazolam
Description: The time that Cmax was observed for 1-Hydroxymidazolam.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 1.000 [0.50 to 3.00] | 1.000 [0.50 to 1.03]

42. Secondary Outcome: Part A: Terminal Elimination Half-life (T½) for Bupropion
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 24 | 24
Hours | 20.577 (2.6082) | 19.203 (2.6331) | 19.383 (2.6591)

43. Secondary Outcome: Part A: t1/2 6-Hydroxybupropion
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Hours | 26.228 (5.9780) | 23.220 (4.9391) | 21.500 (4.3406)

44. Secondary Outcome: Part A: T1/2 for Repaglinide
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment B | Part A: Period 2: Treatment F
Number analyzed (Participants) | 19 | 25
Hours | 4.684 (1.6568) | 6.242 (1.3469)

45. Secondary Outcome: Part A: T1/2 for Flurbiprofen
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 6.906 (1.2545) | 6.855 (1.2666)

46. Secondary Outcome: Part A: T1/2 for Omeprazole
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 24 | 24
Hours | 0.945 (0.3240) | 0.891 (0.2785)

47. Secondary Outcome: Part A: T1/2 for 5-Hydroxyomeprazole
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 1.455 (0.5103) | 1.387 (0.2029)

48. Secondary Outcome: Part A: T1/2 for Midazolam
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Hours | 4.502 (1.7340) | 5.497 (0.6465)

49. Secondary Outcome: Part A: T1/2 for 1-Hydroxymidazolam
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 23 | 25
Hours | 3.346 (4.0653) | 3.172 (0.9569)

50. Secondary Outcome: Part A: Ratio of Metabolite to Parent AUCt Corrected for Molecular Weight (AUCt M/P) for 6-Hydroxybupropion/Bupropion
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: Period 1 Treatment A | Part A: Period 2: Treatment D | Part A: Period 2: Treatment G
Number analyzed (Participants) | 26 | 25 | 24
Ratio | 12.79 (40) | 10.92 (39) | 15.53 (47)

51. Secondary Outcome: Part A: Ratio of Metabolite to Parent AUCt Corrected for Molecular Weight for 5-Hydroxyomeprazole/Omeprazole
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Ratio | 0.5417 (52) | 0.8096 (60)

52. Secondary Outcome: Part A: Ratio of Metabolite to Parent AUCt Corrected for Molecular Weight for Hydroxymidazolam/Midazolam
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: Period 1: Treatment A | Part A: Period 2: Treatment E
Number analyzed (Participants) | 26 | 25
Ratio | 0.4704 (43) | 0.3638 (26)

53. Secondary Outcome: Part B: Tmax for Metformin
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
Hours | 1.500 [1.00 to 5.00] | 2.000 [1.50 to 4.00]

54. Secondary Outcome: Part B: Tmax for Furosemide
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Groups:
- Part B, Period 1: Treatment A: On Period 1 Day 1, participants were administered single oral doses of metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg (Treatment A).
Arm/Group | Part B, Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
Hours | 0.510 [0.50 to 1.00] | 0.775 [0.50 to 1.50]

55. Secondary Outcome: Part B: Tmax for Rosuvastatin
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
Hours | 5.000 [2.50 to 5.05] | 2.500 [1.50 to 5.02]

56. Secondary Outcome: Part B: T½ for Metformin
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 18 | 18
Hours | 3.554 (0.9523) | 3.324 (0.8515)

57. Secondary Outcome: Part B: T½ for Furosemide
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 15 | 17
Hours | 7.786 (5.1296) | 4.757 (2.1595)

58. Secondary Outcome: Part B: T½ for Rosuvastatin
Description: T½ was calculated as ln (2)/lambda z; where lamda z: apparent terminal elimination rate constant.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part B: Period 1: Treatment A | Part B: Period 2: Treatment C
Number analyzed (Participants) | 17 | 18
Hours | 11.436 (8.9813) | 8.852 (3.1587)

59. Other Pre Specified Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. TEAE: any event that was not present before exposure to study drug (voxelotor or cocktail drugs [probe substrates]) or any event already present that worsened in either intensity or frequency after exposure to study drug. An SAE was defined as an AE that at any dose resulted in any of the following outcomes: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability; a congenital anomaly/birth defect; other important medical events.
Time Frame: From start of study drug on Day 1 up to Day 28 (for a maximum of 30 days)
Population: Safety analysis set (SAS) included all participants who received any amount of study drug (voxelotor or cocktail drugs [probe substrates]). As prespecified in the statistical analysis plan, safety data is reported period-wise.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Period 1: On Day 1 of Period 1, participants were administered a single oral dose of Treatment A (bupropion 150 mg, flurbiprofen 50 mg, omeprazole 20 mg, and midazolam 2 mg) and on Day 4, participants received a single oral dose of repaglinide 0.5 mg (Treatment B). Period 1 for Part A was of 5 days.
- Part A: Period 2: In Period 2, participants were administered once daily oral dose of voxelotor 1500 mg (Treatment C) for 13 days. On Day 2, a single oral dose of bupropion 150 mg (Treatment D) was administered immediately following voxelotor administration. On Day 4, single oral dose of Treatment E (flurbiprofen 50 mg, omeprazole 20 mg and midazolam 2 mg) was administered immediately following voxelotor administration. Participants received Treatment F (single oral dose of repaglinide 0.5 mg) and Treatment G (single oral dose of bupropion 150 mg) on Day 6 and Day 12, immediately following voxelotor administration. Period 2 for Part A was of 15 days. There was a washout period of 7 to 14 days in between Period 1 and 2. Participants had a follow-up visit on Day 28.
Arm/Group | Part A: Period 1 | Part A: Period 2
Number analyzed (Participants) | 26 | 25
Participants
  TEAEs | 4 | 9
  SAEs | 0 | 0

60. Other Pre Specified Outcome: Part B: Number of Participants With TEAEs and SAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. TEAE: any event that was not present before exposure to study drug (voxelotor or cocktail drugs [probe substrates]) or any event already present that worsened in either intensity or frequency after exposure to study drug. An SAE was defined as an AE that at any dose resulted in any of the following outcomes: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability; a congenital anomaly/birth defect; other important medical events.
Time Frame: From start of study drug on Day 1 up to Day 18 (for a maximum of 20 days)
Population: SAS included all participants who received any amount of study drug (voxelotor or cocktail drugs [probe substrates]). As prespecified in the statistical analysis plan, safety data is reported period-wise.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Period 1: On Day 1 of Period 1, participants were administered a single oral dose of Treatment A (metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg). Period 1 for Part B was of 4 days.
- Part B: Period 2: In Period 2, from Day 1 to Day 3, participants were administered Treatment B (oral doses of voxelotor 1500 mg) orally for 3 days. On Day 4, participants were administered Treatment C (single oral doses of metformin 10 mg, furosemide 1 mg, and rosuvastatin 10 mg) immediately following voxelotor administration. On Day 5, participants were administered Treatment D (single oral dose of voxelotor 1500 mg). Period 2 for Part B was of 7 days. There was a washout period of 7 to 14 days in between Period 1 and 2. Participants had a follow-up visit on Day 18.
Arm/Group | Part B: Period 1 | Part B: Period 2
Number analyzed (Participants) | 18 | 18
Participants
  TEAEs | 1 | 2
  SAEs | 0 | 0

61. Other Pre Specified Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests
Description: The following laboratory parameters were assessed: hematology: hematocrit, hemoglobin, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, red blood cell count, neutrophils, monocytes, lymphocytes, basophils and eosinophils. coagulation: prothrombin time, partial thromboplastin time, international normalized ratio. Serum Chemistry: albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, creatinine, blood urea nitrogen, lactate dehydrogenase. Urinalysis: ketones, pH, protein, blood glucose, bilirubin, chloride, bicarbonate, phosphorous, potassium was assessed. Clinical significance of laboratory abnormalities was determined by investigator.
Time Frame: From start of study drug on Day 1 up to Day 28 (for a maximum of 30 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Period 1 | Part A: Period 2
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

62. Other Pre Specified Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Physical Examinations
Description: A complete physical examination included cardiovascular, respiratory, gastrointestinal, and neurological systems. Height and weight were also measured and recorded. Clinical significance of physical examinations was determined by investigator.
Time Frame: From start of study drug on Day 1 up to Day 28 (for a maximum of 30 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Period 1 | Part A: Period 2
Number analyzed (Participants) | 26 | 25
Participants | 1 | 0

63. Other Pre Specified Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included oral temperature, heart rate, respiratory rate (breaths per minute), and blood pressure. Blood pressure and heart rate were measured in a supine position using completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Clinical significance of vital signs was determined by investigator.
Time Frame: From start of study drug on Day 1 up to Day 28 (for a maximum of 30 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Period 1 | Part A: Period 2
Number analyzed (Participants) | 26 | 25
Participants | 0 | 1

64. Other Pre Specified Outcome: Part B: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests
Description: as for outcome 61
Time Frame: From start of study drug on Day 1 up to Day 18 (for a maximum of 20 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Period 1 | Part B: Period 2
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

65. Other Pre Specified Outcome: Part B: Number of Participants With Clinically Significant Abnormalities in Physical Examinations
Description: as for outcome 62
Time Frame: From start of study drug on Day 1 up to Day 18 (for a maximum of 20 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Period 1 | Part B: Period 2
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

66. Other Pre Specified Outcome: Part B: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: as for outcome 63
Time Frame: From start of study drug on Day 1 up to Day 18 (for a maximum of 20 days)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Period 1 | Part B: Period 2
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: from start of study drug on Day 1 up to Day 28 (for a maximum of 30 days). Part B: from start of study drug on Day 1 up to Day 18 (for a maximum of 20 days)
Description: Safety population included all participants who received any amount of study drug (voxelotor or cocktail drugs [probe substrates]). As prespecified in the statistical analysis plan, safety data is reported period-wise.
Arm/Group | Part A: Period 1 | Part A: Period 2 | Part B: Period 1 | Part B: Period 2
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/26 | 9/25 | 1/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Period 1 (N=26) | Part A: Period 2 (N=25) | Part B: Period 1 (N=18) | Part B: Period 2 (N=18)
Headache (Nervous system disorders) | 0 | 7 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT05981365/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT05981365/SAP_001.pdf